CLINICAL TRIAL: NCT04423341
Title: Effect of Non-psychoactive Cannabidiol as an Adjunct to Botulinum Toxin in Blepharospasm - a Prospective Double-masked Cross-over Study
Brief Title: Effect of Non-psychoactive Cannabidiol as an Adjunct to Botulinum Toxin in Blepharospasm
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Silkiss Eye Surgery (Other)
Collaborators: Benign Essential Blepharospasm Research Foundation (Other); GW Pharmaceuticals Ltd (Industry); Smith-Kettlewell Eye Research Institute (Other)
Responsible Party: Principal Investigator, Rona Silkiss, MD FACS, Physician, Silkiss Eye Surgery
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1268646
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Blepharospasm; Blepharospasm, Benign Essential; CBD
Keywords: Cannabidiol; Epidiolex; Botulinum Toxin; Eyeblink analysis; Videorecording; Blepharospasm; BEB
MeSH Terms: conditions — Blepharospasm; Benign essential blepharospasm | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A - active medication followed by placebo (Active Comparator)
  Interventions: Drug: Cannabidiol Oral Solution [Epidiolex]
- Group B - placebo followed by active medication (Active Comparator)
  Interventions: Drug: Cannabidiol Oral Solution [Epidiolex]

INTERVENTIONS:
Drug: Cannabidiol Oral Solution [Epidiolex] — 100 mg BID for three months Placebo oral solution for three months

SUMMARY:
The planned study is a prospective analysis of non-psychoactive Cannabidiol (without THC) as an adjunctive therapy for blepharospasm in a masked double cross-over study. This prospective study is a follow-up to a retrospective study completed by the researchers using over-the-counter, self purchased CBD. This study will use FDA approved Cannabidiol medication, Epidiolex, directly from GW pharmaceuticals, rather than self-purchased CBD from the internet. Patients will undergo videorecording with a high resolution videocamera system at days 0, 45, 90, 135, and 180 using a novel blink analysis to gather objective data measurements of changes induced by CBD in Blepharospasm patients. This study will attempt to codify the data and quantify if adjunctive CBD therapy improves those areas compared to botulinum injection alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the private practice of the principal investigator with an ICD code of "blepharospasm" and:
* undergoing routine maximal botulinum therapy
* experiencing break through symptoms of spasm
* marijuana naïve

Exclusion Criteria:

* concomitant diagnosis of epilepsy
* patients whom are not marijuana naive
* patients on concurrent anti-epileptics
* patients who are pregnant or wishing to become pregnant
* patients not wishing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Eyeblink analysis from high speed videocamera recordings - see separate outcome measures | 4 measurements over 6 months
  All patients will undergo video recording of their eyelid kinematics at days 0, 45, 90, 135, and 180. A high-resolution commercially available video camera will capture the eyelid positions at a sampling rate of thirty frames per second. Patients will be assessed in three different lighting conditions - in regular exam room lighting, under examination with the glare source of an indirect ophthalmoscope (at 2000 lux on both eyes from 5 feet), and in dim lighting. The upper and lower eyelid positions captured from each frame of the videos will be input into custom software developed by Visage Technologies, which fits a feature template to the facial features in each frame, including the upper and lower lids of each eye. The difference between the upper and lower lid positions defined the lid aperture, also known as the palpebral fissure. The eyeblink parameters will then calculated from the eyelid aperture time series with custom software written in MATLAB.
Median Blink Amplitude | 4 measurements over 6 months
  Measured in millimeters (mm)

SECONDARY OUTCOMES:
Median Blink Duration | 4 measurements over 6 months
  Measured in milliseconds (ms)
Median Max Blink Velocity | 4 measurements over 6 months
  Measured in millimeters per milliseconds (mm/ms)
Number of Blinks per 100ms | 4 measurements over 6 months
  Total "blinks" in 100 milliseconds (numeric value)

CONTACTS AND LOCATIONS:
Locations (1):
- Silkiss Eye Surgery, Oakland, California, United States

REFERENCES:
- [Derived] Silkiss RZ, Koppinger J, Truong T, Gibson D, Tyler C. Cannabidiol as an Adjunct to Botulinum Toxin in Blepharospasm - A Randomized Pilot Study. Transl Vis Sci Technol. 2023 Aug 1;12(8):17. doi: 10.1167/tvst.12.8.17. PMID 37606606